CLINICAL TRIAL: NCT00363974
Title: An Open-Label Phase I/II Study of XIAP Antisense AEG35156 Administered to Patients With Refractory/Relapsed AML in Combination With Chemotherapy
Brief Title: Study of XIAP Antisense Given With Chemotherapy for Refractory/Relapsed AML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aegera Therapeutics (Industry)
Responsible Party: Jacques Jolivet, MD, Senior VP Clinical, Aegera Therapeutics Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEG35156-103; MDA 2005-0384; PMH 05-0452-C
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Leukemia, Myelomonocytic, Acute
Keywords: AML; leukemia; relapse; refractory; antisense; oligonucleotide
MeSH Terms: conditions — Leukemia, Myelomonocytic, Acute; Leukemia; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: XIAP antisense — 2 days loading dose followed by weekly 2hr infusion

SUMMARY:
The purpose of this study is to determine if the drug, called AEG35156, can be safely given to AML patients and whether it effectively reduces levels of a protein (XIAP) to increase the sensitivity of cancer cells to chemotherapy (ara-C and idarubicin) in patients with refractory or relapsed AML.

DETAILED DESCRIPTION:
This is a phase I/II, single-arm, open-label, study to establish the recommended dose and activity of AEG35156 administered as a daily x3 two-hour infusion prior to reinduction chemotherapy with idarubicin and ara-C followed by weekly two-hour AEG35156 infusions. Subjects eligible for study entry must have confirmed diagnosis of AML in first relapse after an initial CR that lasted less than 6 months or primary refractory AML. Fixed dose of idarubicin and ara-C will be given, plus one of eight doses of AEG35156: 12, 24, 48, 75, 110, 165, 250 and 350mg/m2. A maximum of 54 patients will be treated in cohorts of size 3, starting at 12mg/m2, and not skipping any untried dose level when escalating. Following dose escalation, approximately 20 patients will be treated at the best acceptable dose as determined by the method of Thall and Cook (2004).

ELIGIBILITY:
Inclusion Criteria

* Subjects with relapsed or refractory AML, except those with APL (acute promyelocytic leukemia), that are about to receive their initial treatment for first relapse after an initial CR that lasted less than 6 months or for primary refractory AML that have an expected complete response rate ≤20%. The initial diagnosis of AML has to be based on the presence of > 10% blasts in marrow or blood, and the diagnosis of relapsed/refractory AML based on the presence of either > 10% blasts in marrow or blood or 5-10% blasts in either site together with cytopenia (Hb < 10 g/dL, or platelets < 100,000 /uL, or neutrophil count < 1000 /uL).
* Peripheral AML blast count < 50,000 /uL that is not projected to rise above 50,000 /uL within 5 days of beginning treatment.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Subjects must be >18 years old.
* Male, or female subjects who are post-menopausal (amenorrhagic for at least 12 months), or surgically or biologically sterile. Females of childbearing potential with a negative serum pregnancy test 72-96 hours prior to the 1st infusion in the study and using adequate forms of contraception for the duration of the study, including 30 days after the last treatment. Adequate methods of contraception should be used by both male and female subjects.
* Subjects must have adequate organ and immune function as indicated by the following laboratory values:

  * Parameter Laboratory Values
  * Serum creatinine; <2.0mg/dL
  * Total Bilirubin <2.0mg/dL
  * AST (SGOT) and ALT (SGPT) <3 X ULN * *ULN: Institution's upper limit of normal.
* The subject must understand and be able and willing and likely to fully comply with study procedures, including scheduled follow-up, and restrictions.
* The subject, or the subject's legal guardian, must have given written personally signed and dated informed consent to participate in the study, in accordance with the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guidelines, before completing any study related procedures.

Exclusion Criteria

* Clinical evidence of active CNS leukemic involvement.
* Patients with left-ventricular ejection fractions <50%.
* Active and uncontrolled infection. Patients with an infection that are under active treatment with antibiotics and whose infections are controlled may be entered to the study.
* Current evidence of invasive fungal infection (blood or tissue culture).
* Current evidence of an active second malignancy except for non-melanoma skin cancer.
* Uncontrolled medical problems, unrelated to the malignancy, or of sufficient severity that in the opinion of the investigator, impair a subject's ability to give informed consent or unacceptably reduce the safety of the proposed treatment.
* Neurological or psychiatric disorders that would interfere with consent or study follow-up.
* Known or suspected intolerance or hypersensitivity to the study materials [or closely related compounds] or any of their stated ingredients.
* History of alcohol or other substance abuse within the last year.
* Use of another investigational agent or participation in a clinical trial within the last 14 days prior to enrolment. Subjects who have used a previous AS agent for at least 90 days will be excluded.
* Female subjects who are pregnant or lactating, or females with a positive pregnancy test at screening must be excluded.
* Subjects that have previously been enrolled into this study and subsequently withdrawn must also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2005-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Dose at which AEG35156 when combined with fixed doses of ara-C and idarubicin, produces acceptable CR and toxicity rates as defined and observed at 30 days post-last dose | 1 year

SECONDARY OUTCOMES:
Effects of AEG35156 on XIAP mRNA and protein expression and plasma pharmacokinetic profile of AEG35156. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Jolivet, MD, Study Director — Aegera Therapeutics Inc.
Locations (7):
- United States (5):
  - Norris Cancer Center - University of Southern California, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Johns Hopkins - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - M.D. Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec

REFERENCES:
- [Background] Thall PF, Cook JD. Dose-finding based on efficacy-toxicity trade-offs. Biometrics. 2004 Sep;60(3):684-93. doi: 10.1111/j.0006-341X.2004.00218.x. PMID 15339291